CLINICAL TRIAL: NCT05909969
Title: Development and Validation of the Pelvi-Fit App for Women With Urinary Incontinence.
Brief Title: Development and Validation of Pelvi-Fit App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Yusra Niazi
Record Dates: First submitted 2023-06-11; First posted 2023-06-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: This will be a Pretest-Postest Design with parallel assignment of patients into two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvi-Fit Group (Experimental): The experiment group will receive the treatment protocol for urinary incontinence based on evidence-based protocol through the Pelvi-Fit app.
  Interventions: Other: Pelvi-Fit app Training
- Control (Other): This group will receive the same treatment protocol in a descriptive form (non-app-based treatment) for urinary incontinence.
  Interventions: Other: Control

INTERVENTIONS:
Other: Pelvi-Fit app Training — This group will receive Pelvic Floor Muscle Strengthening exercises through software application.
  Arms: Pelvi-Fit Group
Other: Control — This group will receive Pelvic Floor Muscle Strengthening exercises through instructions and pamphlets describing exercises.
  Arms: Control

SUMMARY:
Urinary incontinence (UI) is defined as involuntary urinary leakage or inability to control urine. Various physiological changes during pregnancy, including collagen changes, hormonal changes, and increased uterine and fetal weight, contribute to the weakening of the pelvic floor muscles (PFMs) during pregnancy. Approximately, 42% of women experience their first UI during pregnancy, and up to 31% of parous women have UI. Women with persistent UI after delivery may continue to experience UI for another 12 years. Therefore, UI during pregnancy may be an essential risk factor for subsequent UI among women. This Study will result in a product called Pelvi-Fit app that will help patients to self-treat their Pelvic Floor disorders in a way that is approved by medical experts. It will allow the patient to train their pelvic floor muscles independently who are not able to get medical assistance due to being in remote areas or any other reason.

DETAILED DESCRIPTION:
Literature suggests that UI is troublesome, affects women's quality of life physically, emotionally, spiritually, and financially. Those who experience it may resort to various methods to deal with the problem, including using pads or incontinence diapers and avoiding social situations because of embarrassment. However, many women do not seek help despite having UI symptoms because of the perception of UI as embarrassment to initiate a discussion about UI with their health care provider. Some are unaware of treatment availability, such as PFM training (PFMT), whereas others feel they should not disturb their health care provider as UI is a temporary issue. Developing a positive attitude is essential to enable people to change their behavior successfully. The use of persuasive technology (PT) in mHealth apps may support attitude and behavior change in users to adopt PFMT as part of their lifestyle. The pre-final version of Pevi-Fit app will be made in this study. The control group will receive the validated content-based treatment protocol of UI in descriptive form and the experiment group will receive the same treatment of UI through pre-final version of the Pelvi-Fit app. The results of both groups will be recorded and compared to assess the effectiveness of using technological methods in the treatment of patients with Urinary Incontinence

ELIGIBILITY:
Inclusion Criteria:

* Females of child-bearing age up to 65 years of age having Urinary Incontinence.
* Females having Cognitive ability to use the Pelvi-Fit App, screened through MMSE tool (Average score >25).

Exclusion Criteria

* Patients of neurological conditions; SCI, Stroke.
* Not friendly to use mobile apps.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incontinence Severity Index | Changes from Baseline to 8th week
  The severity index is based on information about frequency (four levels) and amount of leakage (two or three levels). By multiplication, an index value (1-8 or 1-12) is reached. This index value is further categorized into a severity index of three or four levels.
ICIQ-UI SF- Questionnaire | Changes from Baseline to 8th week
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) evaluates the severity of UI symptoms and their impact on health-related quality of life. When using the ICIQ-UI SF, a total ICIQ score with a range from 0-21 is achieved from the first three questions. The (ICIQ-UISF) is a brief and psychometrically robust patient-completed questionnaire for evaluating the frequency, severity and impact on quality of life (Qu) of urinary incontinence in men and women in research and clinical practice across the world. It is scored on a scale from 0-21.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD, Principal Investigator — Riphah International University
Locations (1):
- Al-Hussain Miternity Clinic, Mianwali, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bi X, Zhao J, Zhao L, Liu Z, Zhang J, Sun D, Song L, Xia Y. Pelvic floor muscle exercise for chronic low back pain. J Int Med Res. 2013 Feb;41(1):146-52. doi: 10.1177/0300060513475383. Epub 2013 Jan 23. PMID 23569140
- [Background] Pedraza R, Nieto J, Ibarra S, Haas EM. Pelvic muscle rehabilitation: a standardized protocol for pelvic floor dysfunction. Adv Urol. 2014;2014:487436. doi: 10.1155/2014/487436. Epub 2014 Jun 11. PMID 25006337
- [Background] Garcia-Sanchez E, Avila-Gandia V, Lopez-Roman J, Martinez-Rodriguez A, Rubio-Arias JA. What Pelvic Floor Muscle Training Load is Optimal in Minimizing Urine Loss in Women with Stress Urinary Incontinence? A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Nov 8;16(22):4358. doi: 10.3390/ijerph16224358. PMID 31717291
- [Background] Jacomo RH, Nascimento TR, Lucena da Siva M, Salata MC, Alves AT, da Cruz PRC, Batista de Sousa J. Exercise regimens other than pelvic floor muscle training cannot increase pelvic muscle strength-a systematic review. J Bodyw Mov Ther. 2020 Oct;24(4):568-574. doi: 10.1016/j.jbmt.2020.08.005. Epub 2020 Sep 10. PMID 33218562
- [Background] Gluppe SB, Engh ME, Bo K. Immediate Effect of Abdominal and Pelvic Floor Muscle Exercises on Interrecti Distance in Women With Diastasis Recti Abdominis Who Were Parous. Phys Ther. 2020 Aug 12;100(8):1372-1383. doi: 10.1093/ptj/pzaa070. PMID 32302393
- [Background] Jaffar A, Tan CE, Mohd-Sidik S, Admodisastro N, Goodyear-Smith F. Persuasive Technology in an mHealth App Designed for Pelvic Floor Muscle Training Among Women: Systematic Review. JMIR Mhealth Uhealth. 2022 Mar 22;10(3):e28751. doi: 10.2196/28751. PMID 35315777
- [Background] Widdison R, Rashidi A, Whitehead L. Effectiveness of mobile apps to improve urinary incontinence: a systematic review of randomised controlled trials. BMC Nurs. 2022 Jan 28;21(1):32. doi: 10.1186/s12912-022-00812-6. PMID 35090464
- [Background] Gron Jensen LC, Boie S, Axelsen S. International consultation on incontinence questionnaire - Urinary incontinence short form ICIQ-UI SF: Validation of its use in a Danish speaking population of municipal employees. PLoS One. 2022 Apr 6;17(4):e0266479. doi: 10.1371/journal.pone.0266479. eCollection 2022. PMID 35385519
- [Derived] Niazi YM, Riaz H, Naeem M, Saeed A. Development of the Pelvi-Fit app for women with urinary incontinence. Eur J Obstet Gynecol Reprod Biol. 2025 Dec;315:114726. doi: 10.1016/j.ejogrb.2025.114726. Epub 2025 Sep 17. PMID 40997686